CLINICAL TRIAL: NCT04609189
Title: Pearlium®/Effecti-Cal®, a Novel Formulation of Calcium, Vitamin D and Minerals for Prevention of Postmenopausal Bone Loss
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pro00020853
Record Dates: First submitted 2020-10-23; First posted 2020-10-30 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2020-10

CONDITIONS: Osteoporosis, Postmenopausal
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Calcium Carbonate; Cholecalciferol

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pearlium®/EffectiCal® (Experimental)
  Interventions: Drug: Pearlium/EffectiCal
- Calcium Carbonate/Vitamin D3 (Active Comparator)
  Interventions: Drug: Calcium carbonate/vitamin D3

INTERVENTIONS:
Drug: Pearlium/EffectiCal — Oral administration of Pearlium/EffectiCal.
  Arms: Pearlium®/EffectiCal®
Drug: Calcium carbonate/vitamin D3 — Oral administration of Calcium Carbonate/Vitamin D3
  Arms: Calcium Carbonate/Vitamin D3

SUMMARY:
Postmenopausal osteoporosis is one of the important medical disorders affecting women after menopause. It is characterized by bone loss and reduced bone strength. In turn, this leads to increased risk of fracture. Bone loss in postmenopausal women occurs when calcium leaks out of the bones. Supplementing calcium and vitamin D is considered as standard prophylactic measures against osteoporosis for postmenopausal women over age 50.

Currently, various formulations of calcium salt are under development for the effective supplementation of calcium. Pearlium/Effecti-Cal is a new formulation optimized for high solubility of calcium salt. Formulation A5 (the base formulation of Pearlium/Effecti-Cal) showed three fold higher retention of calcium in rats than calcium carbonate (the most popular calcium supplement). High retention of calcium allowed the reduction of orally administered calcium for the same effect. This can contribute to the reduction of gastrointestinal side effects such as constipation.

In postmenopausal women, bone mineral loss is reflected on the elevated level of bone turnover markers. In this study, the efficacy of Pearlium/Effecti-Cal will be assessed by the suppression of bone turnover markers. In addition, the safety of Pearlium/Effecti-Cal will be evaluated with a bowel function diary, which can capture the profile of constipation symptoms.

The participants will experience run-in period (two months) for removing the residual effect of previously taken health product on bone turnover. For the following treatment period (six months), one hundred and two participants will be allocated by chance into groups for the treatment of Pearlium/Effecti-Cal or active comparator (conventional calcium supplement).

ELIGIBILITY:
Inclusion Criteria:

1. Female of age 40 to 85, inclusive
2. Have been postmenopausal for at least 3 years. Menopause is defined by a history of amenorrhea for at least 12 consecutive months since the end of the final menstrual period and plasma Follicle-stimulating hormone > 30 IU/L. In the case of hysterectomy, the date of the surgery is regarded as the end of the final menstrual period. Postmenopausal period is calculated from the end of the final menstrual period.
3. Ambulatory
4. Competent and willing to give signed informed consent

Exclusion Criteria:

1. Health conditions or any history that can invalidate the evaluation of bone mineral density (BMD) by dual energy x-ray absorptiometry
2. The lowest T-score in dual energy x-ray absorptiometry report less than the age-specific limit of T-score
3. A history of bilateral oophorectomy before age 40
4. A history of menopause before age 40
5. A history of malignancy within the past 3 years, except basal cell carcinoma of the skin
6. Current history of any medical disease that may be associated with the development of metabolic bone disease
7. Body Mass Index (BMI) < 18.5 kg/m2 or > 38.0 kg/m2 at the screening visit
8. Vigorous physical activities for more than 180 minutes/week
9. Any screening laboratory abnormality that exceeds the local laboratory's reference range by more than Investigators pre-specified limits
10. Use of medications or supplements which can affect bone or calcium metabolism
11. Use of any other investigational drugs during the past 1 month
12. Clinically significant and currently active hematological, endocrinological, cardiovascular, renal, hepatic, gastrointestinal psychiatric or neurological conditions.
13. Any other medical condition or reason that, in the Investigator's opinion, makes the participant unsuitable for this study
14. Mental incapacity or language barriers which preclude adequate understanding or cooperation
15. Unwillingness to comply with the requirements of the study protocol

Ages: 40 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Actual)
Dates: Start 2012-07-12 (Actual); Primary Completion 2014-05-02 (Actual); Study Completion 2014-05-02 (Actual)

PRIMARY OUTCOMES:
Percentage change from baseline in bone turnover markers | Baseline to Week 34
  Percentage change from baseline in bone turnover markers (C-telopeptide of type I collagen (CTx) and N-terminal propeptide of type I collagen (PINP))

SECONDARY OUTCOMES:
Vitamin D levels | Baseline to Week 34
  Percent change in the 25-hydroxy vitamin D3 levels in blood
Parathyroid hormone levels | Baseline to Week 34
  Percent change in parathyroid levels in blood
Constipation profile - Comparisons of strain for each bowel movement in 14-day assessment | Baseline to Week 34
  Constipation will be monitored with the bowel function diary. This diary assesses the symptoms related with bowel movements, and collects information on the frequency of the bowel movements. The minimum value is 1 and the maximum value is 5, a higher score indicates a worse outcome.
Constipation profile - Comparisons of ability to fully empty bowels for each bowel movement in 14-day assessment | Baseline to Week 34
  Constipation will be monitored with the bowel function diary. This diary assesses the symptoms related with bowel movements, and collects information on the frequency of the bowel movements. The minimum value is 1 and the maximum value is 5, a higher source indicates a better outcome.
Constipation profile - Comparisons of pain around rectum for each bowel movement in 14-day assessment | Baseline to Week 34
  Constipation will be monitored with the bowel function diary. This diary assesses the symptoms related with bowel movements, and collects information on the frequency of the bowel movements. The minimum value is 1 and the maximum value is 5, a higher score indicates a worse outcome.
Constipation profile - Comparisons of Bristol Stool score for each bowel movement in 14-day assessment | Baseline to Week 34
  Consistency of bowel movements will assessed using the Bristol Stool score. The minimum value is 1 and the maximum value is 7, a higher score indicates a better outcome.
Constipation profile - Comparisons of time of each bowel movement in a day in 14-day assessment | Baseline to Week 34
  Assessed from the bowel function diary.
Constipation profile - Comparisons of inability to have a bowel movement in 24-hours assessment in 14-day period | Baseline to Week 34
  Constipation will be monitored with the bowel function diary. This diary assesses the symptoms related with bowel movements, and collects information on the frequency of the bowel movements. The minimum value is 1 and the maximum value is 5, a higher score indicates a worse outcome.
Constipation profile - Comparisons of bloating in 24-hours assessment of bowel movements in 14-day period | Baseline to Week 34
  Constipation will be monitored with the bowel function diary. This diary assesses the symptoms related with bowel movements, and collects information on the frequency of the bowel movements. The minimum value is 1 and the maximum value is 6, a higher score indicates a worse outcome.
Constipation profile - Comparisons of pain in abdomen in 24-hours assessment of bowel movements in 14-day period | Baseline to Week 34
  Constipation will be monitored with the bowel function diary. This diary assesses the symptoms related with bowel movements, and collects information on the frequency of the bowel movements. The minimum value is 1 and the maximum value is 6, a higher score indicates a worse outcome.
Constipation profile - Comparisons of botheration by gas in 24-hours assessment of bowel movements in 14-day per | Baseline to Week 34
  Constipation will be monitored with the bowel function diary. This diary assesses the symptoms related with bowel movements, and collects information on the frequency of the bowel movements. The minimum value is 1 and the maximum value is 6, a higher score indicates a worse outcome.
Constipation profile - Comparisons of lack of appetite in 24-hours assessment of bowel movements in 14-day period | Baseline to Week 34
  Constipation will be monitored with the bowel function diary. This diary assesses the symptoms related with bowel movements, and collects information on the frequency of the bowel movements. The minimum value is 1 and the maximum value is 5, a higher score indicates a worse outcome.